CLINICAL TRIAL: NCT05644145
Title: Estudio Sobre Respuesta de Anticuerpos Neutralizantes Contra la Fiebre Amarilla Cuatro a Siete años después de Vacunar Una población pediátrica Entre Los 12 y 23 Meses de Edad en Argentina
Brief Title: Immunogenicity of Yellow Fever Vaccine in a Pediatric Population Vaccinated at 12-23 Months of Age in Argentina
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Public Health, Argentina (Other Government)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Pan American Health Organization (Other)
Responsible Party: Principal Investigator, Andrea Uboldi, medico pediatra infectologo, Ministry of Public Health, Argentina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IS003815
Record Dates: First submitted 2022-11-11; First posted 2022-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Yellow Fever
Keywords: Antibodies response; Yellow Fever Vaccine
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Intervention Model Description: It is a seroepidemiological study to evaluate the Immunization Program. It is a serological survey of the cohort of children who participated in the preliminary investigation and seroconverted after vaccination against yellow fever.
Masking Description: Each enrolled participant is coded, and whoever processes the sample does not know the identity of the children included
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yellow fever seropositive vaccinated pediatric population in Argentina (Experimental): Yellow fever seropositive pediatric population in Argentina after receiving the YF vaccine at 12-23 months of age.
  Interventions: Biological: Serological study after yellow fever vaccination

INTERVENTIONS:
Biological: Serological study after yellow fever vaccination — It is a serological survey of the cohort of children who participated in the preliminary investigation and seroconverted after vaccination against yellow fever.
  Other Names: Immunogenicity after yellow fever vaccine

SUMMARY:
Northern Argentina is a risk area for yellow fever (YF). Recent studies have suggested that immunity wanes in children vaccinated between 9 and 23 months of age. In 2015, a collaborative study conducted by the Ministry of Health (MoH) of Argentina, the Pan American Health Organization (PAHO), and the US Centers for Disease Control and Prevention (CDC) assessed the immunogenicity and safety of co-administration of YF and MMR vaccines in a pediatric population at 12-13 months of age. A total of 741 children presenting for routine immunization at 12-13 months of age enrolled and completed the study. It is now four to seven years since this pediatric group received their YF vaccinations. This cohort is unique because their initial YF vaccination and immune response to the vaccine dose are well characterized. Contact information collected during the earlier study will be used to locate the children. If consent is obtained, a 5ml specimen of blood will be collected and shipped to the CDC's Arboviral Diseases Reference Laboratory (ADRL) in Fort Collins, CO for plaque reduction neutralization testing using a 50% cut-off (PRNT50) to detect YF virus-specific neutralizing antibodies. Children with neutralizing antibody titers that are higher than their baseline titer collected approximately 28 days following YF vaccination will have PRNTs done for cross-reacting flaviviruses.

DETAILED DESCRIPTION:
Yellow fever (YF) continues to be a public health problem for 13 countries in the Americas, including northern Argentina. From 1960 to 2019, these countries reported 9,673 confirmed cases and 2,480 deaths. In the same period, Argentina reported 69 confirmed cases with two deaths. Vaccination against YF is recommended for all children living in risk areas in the Americas. In Argentina, the vaccine was administered at the same visit as the measles, mumps, and rubella (MMR) vaccine at 12 months of age.

A study published in 2011 found that simultaneous vaccination with YF and MMR vaccines had a negative impact on YF, mumps, and rubella seroconversion rates in Brazilian children aged 12 to 23 months. In 2013, the Strategic Advisory Group of Experts (SAGE) on immunization reviewed the available data on the co-administration of the YF vaccine with other inactivated and lived attenuated vaccines. In its June 2013 position paper, the WHO states that the YF vaccine can be co-administered with other vaccines but recommends further studies on co-administration with other vaccines, including MMR. In 2013, the Ministry of Health of Argentina changed the indication age for the YF vaccine to be administered to the pediatric population of 18 months, given concerns about a possible interference with MMR and the number of additional vaccines recommended for the pediatric population of 12 months.

In 2015, a collaborative study between the Ministry of Health (MoH) of Argentina, the Pan American Health Organization (PAHO), and the US Centers for Disease Control and Prevention (CDC) was initiated to assess the immunogenicity and the safety of joint administration of the YF and MMR vaccines in the pediatric population vaccinated at 12-13 months of age. 741 children presenting for routine immunization at 12-13 months of age enrolled and completed the study. Three randomized groups received the YF and MMR vaccines simultaneously or 28 days apart. The study found high seroconversion rates against all antigens in the co-administered and sequential groups. However, the magnitude of the antibody response was lower for YF, rubella, and mumps when the vaccines were co-administered.

The WHO currently states that a single dose of the YF vaccine is sufficient to confer lifelong sustained protective immunity against the disease; a booster dose is unnecessary. However, since the booster dose requirement was removed in 2013, new data have been published from pediatric population cohorts in Brazil, Mali, and Ghana, indicating a decrease in the proportion of children seropositive for neutralizing antibodies over time. Seropositivity rates as low as 28% for children in Ghana have been reported two years after vaccination. Given these findings, WHO and PAHO have prioritized obtaining additional longer-term immunogenicity data for the pediatric population vaccinated against YF.

The children who participated in the Argentina YF and MMR vaccination study provide an opportunity to assess whether the Argentine childhood immunization program provides adequate long-term immunity against YF. The last minor enrolled in 2018; It has been four to seven years since this pediatric group received their regular YF vaccinations. This cohort is unique because their initial YF vaccination and immune response to the vaccine dose are well characterized. This program evaluation is necessary to provide Argentina with evidence to inform future changes to its childhood immunization schedule.

Contact information collected during the co-administration study will be used to locate the children who completed the study. If consent is obtained, a 5ml specimen of blood will be collected and shipped to the CDC's Arboviral Diseases Reference Laboratory (ADRL) in Fort Collins, CO for plaque reduction neutralization testing using a 50% cut-off (PRNT50) to detect YF virus-specific neutralizing antibodies. Children with neutralizing antibody titers that are higher than their baseline titer collected approximately 28 days following YF vaccination will have PRNTs done for cross-reacting flaviviruses.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in the 2015 study received one dose of YF vaccine and had documented seroconversion regardless of the
* Healthy child, determined by clinical history
* Availability to perform a single blood draw
* Informed consent signed by the parents.

Exclusion Criteria:

Children in the 2015 study received one dose of the Yellow Fever vaccine and had NO documented seroconversion.

* Children enrolled in the 2015 study received a dose of the Yellow Fever vaccine and had documented seroconversion but, for different reasons, received a booster (minimum interval of one month between doses).
* Children enrolled in the 2015 study received one dose of the Yellow Fever vaccine and had documented seroconversion but developed Yellow Fever
* Children enrolled in the 2015 study received one dose of the Yellow Fever vaccine and had documented seroconversion but are participating in another clinical drug trial of a drug, vaccine, or medical device
* Children enrolled in the 2015 study received a dose of the Yellow Fever vaccine and had documented seroconversion but, for various reasons, are immunocompromised:

Weakened immune function, including HIV infection, primary immunodeficiencies, having received immunosuppressive doses of oral or injectable corticosteroids (or equivalent), having received immunomodulators or chemotherapeutic agents, disease of the thymus, Severe illness/fever (mild illness without fever is not an exclusion criteria)

● Any condition that, in the judgment of study personnel, poses a risk to the health of the participant or interferes with the assessment of response to the vaccine

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 361 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of the pediatric population seropositive for yellow fever ≥ 4 years after yellow fever vaccination at 12-23 months of age in Argentina. | 4-7 years following vaccination
  The proportion of children with detectable neutralizing antibodies 4-7 years following yellow fever vaccination.

SECONDARY OUTCOMES:
To assess the influence of simultaneous administration versus sequential administration 28 days apart of yellow fever and MMR vaccines on yellow fever seropositivity and neutralizing antibody titers four to seven years later. | 4-7 years following vaccination
  In the co-administration study, the target population was randomized into three groups. Group 1 received the yellow fever and MMR vaccines simultaneously, group 2 received the MMR vaccine followed by the yellow fever vaccine 28 days later, and group 3 received the yellow fever vaccine followed by the MMR vaccine 28 days later.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Vizzotti, Study Chair — Ministry of Public Health, Argentina
Locations (3):
- Argentina (3):
  - SAMIC Eldorado Hospital, Eldorado, Misiones Province
  - SAMIC Obera Hospital, Oberá, Misiones Province
  - Favoloro Hospital, Posadas, Misiones Province

IPD SHARING:
Plan to Share IPD: Yes
Deidentified datasets generated in this study, including particular individual data that underlie the results reported in this article after identification, will be available for three years, starting after publication, to researchers who provide a methodologically sound proposal. All variables deemed to be personally identifiable information will be categorized or removed. The study protocol and informed consent forms will be available also.
Supporting Information: Study Protocol, ICF
Time Frame: It will be available for three years, starting after publication.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal. All variables deemed to be personally identifiable information will be categorized or removed. The information will be available from the lead contact upon request.

REFERENCES:
- [Background] Nascimento Silva JR, Camacho LA, Siqueira MM, Freire Mde S, Castro YP, Maia Mde L, Yamamura AM, Martins RM, Leal Mde L; Collaborative Group for the Study of Yellow Fever Vaccines. Mutual interference on the immune response to yellow fever vaccine and a combined vaccine against measles, mumps and rubella. Vaccine. 2011 Aug 26;29(37):6327-34. doi: 10.1016/j.vaccine.2011.05.019. Epub 2011 Jun 2. PMID 21640779
- [Background] de Noronha TG, de Lourdes de Sousa Maia M, Geraldo Leite Ribeiro J, Campos Lemos JA, Maria Barbosa de Lima S, Martins-Filho OA, Campi-Azevedo AC, da Silva Freire M, de Menezes Martins R, Bastos Camacho LA; Collaborative Group for Studies of Yellow Fever Vaccine. Duration of post-vaccination humoral immunity against yellow fever in children. Vaccine. 2019 Nov 15;37(48):7147-7154. doi: 10.1016/j.vaccine.2019.09.051. Epub 2019 Oct 4. PMID 31590934
- [Background] Campi-Azevedo AC, Reis LR, Peruhype-Magalhaes V, Coelho-Dos-Reis JG, Antonelli LR, Fonseca CT, Costa-Pereira C, Souza-Fagundes EM, da Costa-Rocha IA, Mambrini JVM, Lemos JAC, Ribeiro JGL, Caldas IR, Camacho LAB, Maia MLS, de Noronha TG, de Lima SMB, Simoes M, Freire MDS, Martins RM, Homma A, Tauil PL, Vasconcelos PFC, Romano APM, Domingues CM, Teixeira-Carvalho A, Martins-Filho OA. Short-Lived Immunity After 17DD Yellow Fever Single Dose Indicates That Booster Vaccination May Be Required to Guarantee Protective Immunity in Children. Front Immunol. 2019 Sep 26;10:2192. doi: 10.3389/fimmu.2019.02192. eCollection 2019. PMID 31616412
- [Background] Domingo C, Fraissinet J, Ansah PO, Kelly C, Bhat N, Sow SO, Mejia JE. Long-term immunity against yellow fever in children vaccinated during infancy: a longitudinal cohort study. Lancet Infect Dis. 2019 Dec;19(12):1363-1370. doi: 10.1016/S1473-3099(19)30323-8. Epub 2019 Sep 19. PMID 31543249
- [Background] Vaccines and vaccination against yellow fever. WHO position paper -- June 2013. Wkly Epidemiol Rec. 2013 Jul 5;88(27):269-83. No abstract available. English, French. PMID 23909008
- [Background] Who. Vaccines and vaccination against yellow fever: WHO Position Paper, June 2013--recommendations. Vaccine. 2015 Jan 1;33(1):76-7. doi: 10.1016/j.vaccine.2014.05.040. Epub 2014 May 20. PMID 24852721
- See also: PAHO-WHO Member States reports to Health Emergency Information & Risk assessment Unit (HIM) PAHO Health Emergencies Departments, 2022. Data compilation, analysis and report production. — https://ais.paho.org//phip//viz//ed_yellowfever.asp
- See also: Ropero Alba Maria, 2020. Immunogenicity of Co-administered Yellow Fever and Measles, Mumps, and Rubella (MMR) Vaccines — https://clinicaltrials.gov/ct2/show/NCT03368495?cond=Yellow+Fever&cntry=AR&draw=2&rank=1